CLINICAL TRIAL: NCT07397793
Title: Management of Late Presenting Congenital Diaphragmatic Hernia: A Single Center Experience
Brief Title: Management of Late Presenting Congenital Diaphragmatic Hernia .
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jehad Emam Abdelrahman (Other)
Collaborators: Sohag University (Other)
Responsible Party: Sponsor-Investigator, Jehad Emam Abdelrahman, Resident at pediatric surgery department, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med--25-12-8MS
Record Dates: First submitted 2026-01-06; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional non controlled (Other): Interventional
  Interventions: Procedure: MIS and open surgery repair

INTERVENTIONS:
Procedure: MIS and open surgery repair — Laparoscopic, thoracoscopic and laparotomy surgery

SUMMARY:
Diagnosis and different ways of surgical repair of Congenital diaphragmatic hernia

ELIGIBILITY:
Inclusion Criteria:

1. Presentation between age of 1 month till 15 yrs
2. Underwent surgical repair (open or minimally invasive) at the Pediatric Surgery Department, Sohag University.
3. Patient who has complete preoperative and postoperative data

Exclusion Criteria:

* 1. Types of diaphragmatic hernia other than CDH 2. Incomplete clinical or follow-up data. 3. Patients who underwent surgical repair outside the Pediatric Surgery Department, Sohag University

Ages: 30 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Post operative Survival rate | 2 months
  Spontaneous breathing without distress

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided